CLINICAL TRIAL: NCT02838472
Title: Ascorbic Acid Treatment for Patients With Combined Mineralocorticoid and Glucocorticoid Deficiency Secondary to Nicotinamide Nucleotide Transhydrogenase Mutation
Brief Title: Ascorbic Acid Treatment in Congenital Glucocorticoids and Mineralocorticoids Deficiency Due to NNT Mutation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0631-15-HMO
Record Dates: First submitted 2016-07-17; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-06

CONDITIONS: Glucocorticoids Deficiency
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ascorbic Acid — Ascorbic acid administration at a doses of 75-80% of the upper limit of allowance according to IOM
  Other Names: Vitamin C

SUMMARY:
Nicotinamide nucleotide transhydrogenase (NNT) mutations cause glucocorticoid and mineralocorticoid deficiencies through decreased detoxification of reactive oxygen species (ROS) in adrenocortical cells.

Ascorbic acid is well known by its high antioxidant activity due to the neutralization of free radicals and other reactive oxygen species.

Preliminary results of NNT_p.G200S homozygous fibroblasts' treatment with 10 micro molar L-ascorbic acid shows significant improvement in mitochondrial morphology and in ROS content.

The aim of this study is to figure out if ascorbic acid treatment improves the phenotype of NNT patients by reducing ROS in their adrenocortical cells and preventing their apoptosis.

DETAILED DESCRIPTION:
Most cases of familial glucocorticoid and mineralocorticoid deficiency are caused by mutations interrupting steroidogenesis such as 21- hydroxylase deficiency. Recently, nicotinamide nucleotide transhydrogenase (NNT) mutations were found to cause isolated glucocorticoid deficiency or combined mineralocorticoid and glucocorticoid deficiency through decreased detoxification of reactive oxygen species (ROS) in adrenocortical cells.

NNT mutation in mice causes also glucose intolerance. Ascorbic acid is an essential water-soluble vitamin with excellent reducing properties, well known by its high antioxidant activity due to the neutralization of free radicals and other reactive oxygen species. This vitamin acts as the first line of defense during oxidative stress in the human body.

Ascorbic acid treatment for variant disease (e.g. - cancer, type 2 diabetes, anxiety, depression, asthma and cardiovascular diseases) have been meticulously studies with no major adverse effects.

In a previous study, the investigators demonstrated a higher ROS levels, a lower ATP content and a change in mitochondrial morphology in NNT_p.G200S homozygous fibroblasts compared with control fibroblasts.

Preliminary results of NNT_p.G200S homozygous fibroblasts' treatment with 10 micro molar L-ascorbic acid shows significant improvement in mitochondrial morphology and in ROS content.

The aim of this study is to figure out if ascorbic acid treatment improves the phenotype of NNT patients by reducing ROS in their adrenocortical cells and preventing their apoptosis.

During the study NNT_p.G200S homozygous patients (no.-3) will be hospitalised for ACTH and OGTT tests and start ascorbic acid treatment at a doses of 75-80% of the upper limit of allowance according to IOM. ACTH and OGTT will be repeated 6 months later to assess improvement in glucocorticoids production and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* NNT mutation homozygous patients with glucocorticoids deficiency

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
glucocorticoids secretion in response to ACTH test | 1 year
basal ACTH levels | 1 year

SECONDARY OUTCOMES:
insulin and glucose levels in OGTT | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah medical center, Jerusalem, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meimaridou E, Kowalczyk J, Guasti L, Hughes CR, Wagner F, Frommolt P, Nurnberg P, Mann NP, Banerjee R, Saka HN, Chapple JP, King PJ, Clark AJ, Metherell LA. Mutations in NNT encoding nicotinamide nucleotide transhydrogenase cause familial glucocorticoid deficiency. Nat Genet. 2012 May 27;44(7):740-2. doi: 10.1038/ng.2299. PMID 22634753
- [Background] Institute of Medicine (US) Panel on Dietary Antioxidants and Related Compounds. Dietary Reference Intakes for Vitamin C, Vitamin E, Selenium, and Carotenoids. Washington (DC): National Academies Press (US); 2000. Available from http://www.ncbi.nlm.nih.gov/books/NBK225483/ PMID 25077263
- [Result] Weinberg-Shukron A, Abu-Libdeh A, Zhadeh F, Carmel L, Kogot-Levin A, Kamal L, Kanaan M, Zeligson S, Renbaum P, Levy-Lahad E, Zangen D. Combined mineralocorticoid and glucocorticoid deficiency is caused by a novel founder nicotinamide nucleotide transhydrogenase mutation that alters mitochondrial morphology and increases oxidative stress. J Med Genet. 2015 Sep;52(9):636-41. doi: 10.1136/jmedgenet-2015-103078. Epub 2015 Jun 12. PMID 26070314